CLINICAL TRIAL: NCT07224308
Title: Long-Term Efficacy and Duration of MFU-V at Multiple Depths and at 1.5 mm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Levine Center for Plastic Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT10912
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Laxity; Skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Multi-Depth Ultherapy Prime Treatment (Experimental): Participants in this arm will receive a single full-face and neck Ultherapy Prime treatment delivered at multiple depths according to the manufacturer's guidelines for MFU-V energy placement. Energy will be applied using the appropriate transducers for each anatomical depth to target multiple layers of tissue beneath the skin surface. The goal is to stimulate collagen production at varying focal points to enhance lifting, tightening, and overall skin quality.
  Interventions: Device: Ultherapy Prime
- Single-Depth Ultherapy Prime Treatment (1.5 mm) (Experimental): Participants in this arm will receive a single full-face and neck Ultherapy Prime treatment delivered exclusively at the 1.5 mm depth, which is one of the FDA-cleared depths for treatment of the lower face and neck. This protocol evaluates whether single-depth energy delivery can achieve meaningful skin improvement compared with multi-layer treatment.
  Interventions: Device: Ultherapy Prime

INTERVENTIONS:
Device: Ultherapy Prime — Ultherapy Prime is an FDA-cleared micro-focused ultrasound (MFU-V) device used for non-invasive lifting and tightening of the lower face, submentum, neck, brow, and improvement of décolleté lines. It delivers precise ultrasound energy at controlled depths to create thermal coagulation points that stimulate neocollagenesis, promoting new collagen and elastin for improved firmness and visible lifting. The system includes real-time DeepSEE® imaging to visualize tissue layers and ensure accurate energy placement. Ultherapy Prime uses transducers at FDA-cleared depths such as 1.5 mm, 2.0 mm, 3.0 mm, and 4.5 mm. For this study, treatment is delivered at multiple depths or only at 1.5 mm depending on randomization. It is non-surgical, non-ionizing, does not break the skin, and improvement develops gradually as collagen remodels.

SUMMARY:
The goal of this clinical trial is to evaluate the long-term safety and effectiveness of Ultherapy Prime (MFU-V) for improving lines, wrinkles, laxity, and crepiness of the lower face, submentum, and neck. The study will enroll adult male and female subjects aged 25-65 with moderate to severe lower-face and neck skin laxity who are appropriate candidates for non-invasive ultrasound treatment.

The main questions this study aims to answer are:

Does Ultherapy Prime delivered at multiple depths compared to a single-depth (1.5 mm) treatment improve clinical lifting, tightening, and smoothing of the lower face and neck over a 12-month period?

Does treatment with Ultherapy Prime stimulate measurable improvements in collagen-related skin quality, patient satisfaction, and investigator-assessed aesthetic outcomes?

Because the study includes two treatment approaches, researchers will compare a multi-depth MFU-V treatment protocol versus a single-depth (1.5 mm) MFU-V treatment protocol to determine whether multi-depth energy delivery provides superior or longer-lasting clinical improvement.

What Participants Will Do

Participants will:

Attend a total of 5 study visits over 12 months (Screening/Treatment, 1-month, 3-month, 6-month, and 12-month follow-ups).

Undergo a single Ultherapy Prime treatment session at either multiple depths or at the 1.5 mm depth only.

Complete standardized photography, including 2D and 3D images, at all timepoints.

Participate in clinical assessments, including GAIS scoring, cutometer elasticity measurements (if applicable), and investigator- and patient-reported satisfaction scales.

Follow pre-visit requirements, including:

No moisturizers, lotions, or topical products on the treatment area before each visit

No hair in the treatment area (shave the day prior if needed)

Complete questionnaires evaluating satisfaction, comfort, and perceived treatment benefits.

Adhere to follow-up schedules, avoiding elective aesthetic procedures to the lower face, submentum, or neck during the study period.

DETAILED DESCRIPTION:
This study is a prospective, single-center clinical trial designed to evaluate the long-term safety and effectiveness of Ultherapy Prime (MFU-V) for improving lines, wrinkles, and skin laxity of the lower face, submentum, and neck. Ultherapy Prime is an FDA-cleared focused ultrasound device indicated for non-invasive lifting and tightening of the skin under the chin, on the neck, and on the brow, as well as for improving lines and wrinkles of the décolleté. The device delivers precise micro-focused ultrasound energy at controlled depths beneath the skin's surface to stimulate neocollagenesis-the natural production of new collagen that contributes to skin firmness, elasticity, and support.

The objective of this study is to assess clinical outcomes following a single Ultherapy Prime treatment using either a multi-depth protocol or a single-depth protocol at 1.5 mm. The study will enroll 20 adult subjects aged 25 to 65 with moderate to severe laxity or crepiness of the lower face and neck who are appropriate candidates for non-invasive energy-based treatment.

Participants will be randomized to receive Ultherapy Prime at either multiple treatment depths or at the 1.5 mm depth alone. All subjects will undergo standardized 2D and 3D digital photography, clinical assessments, and patient-reported outcome measures over a 12-month follow-up period. Investigator-assessed and patient-reported evaluations-including the Global Aesthetic Improvement Scale (GAIS), cutometer elasticity measurements (if applicable), and satisfaction scales-will be used to assess changes in skin quality, lifting, tightening, and overall aesthetic improvement.

The study includes five visits: a combined Screening/Treatment Visit, and follow-up visits at 1 month, 3 months, 6 months, and 12 months post-treatment. The Screening/Treatment Visit will include informed consent, eligibility confirmation, pregnancy testing if applicable, baseline imaging, and delivery of the assigned Ultherapy Prime treatment. Participants must avoid applying any lotions, moisturizers, or topical products to the treatment area prior to each visit. The treatment area must be free of hair; if shaving is required, participants must shave the day before treatment.

To reduce confounding variables, subjects must refrain from undergoing elective aesthetic procedures involving the lower face, submentum, or neck for the duration of the 12-month study. Safety will be monitored throughout the trial through documentation of adverse events, subject-reported symptoms, and clinical examinations. Because Ultherapy Prime is already FDA-cleared for the anatomical regions being treated, and because treatment involves a single non-invasive procedure, the study is considered minimal risk.

This research will contribute to a deeper understanding of the duration and extent of clinical benefits associated with Ultherapy Prime, as well as whether multi-depth treatment results in greater or longer-lasting improvement compared to treatment at a single depth.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 25 and 65 years of age at the time of screening.

Presence of moderate to severe laxity, fine lines, or crepiness of the lower face, submentum, and/or neck that is appropriate for improvement with non-invasive MFU-V treatment.

Skin condition not advanced enough to require surgical correction.

Willingness to refrain from elective aesthetic procedures involving the face, submentum, or neck for the entire 12-month duration of the study.

Ability and willingness to comply with all study visits, procedures, and follow-up requirements.

Sufficient English language proficiency to understand study instructions and complete questionnaires.

For participants of childbearing potential: negative urine pregnancy test on the day of treatment and willingness to use adequate contraception during the study.

Ability to provide written informed consent.

Exclusion Criteria:

* Male or female subjects between 25 and 65 years of age at the time of screening.

Presence of moderate to severe laxity, fine lines, or crepiness of the lower face, submentum, and/or neck that is appropriate for improvement with non-invasive MFU-V treatment.

Skin condition not advanced enough to require surgical correction.

Willingness to refrain from elective aesthetic procedures involving the face, submentum, or neck for the entire 12-month duration of the study.

Ability and willingness to comply with all study visits, procedures, and follow-up requirements.

Sufficient English language proficiency to understand study instructions and complete questionnaires.

For participants of childbearing potential: negative urine pregnancy test on the day of treatment and willingness to use adequate contraception during the study.

Ability to provide written informed consent.

Exclusion Criteria:

Active systemic or local skin disease (e.g., eczema, psoriasis, dermatitis, infection) that may affect wound healing or the evaluation of results.

Scarring, tattoos, or significant pigmentary alterations in the planned treatment areas.

Metallic implants or other implanted electronic devices (e.g., pacemakers) in or near the treatment area.

Open wounds, lesions, active herpes simplex, or active cystic/severe inflammatory acne in the treatment area.

Use of isotretinoin or other oral retinoids within the past 12 months or planned use during the study.

Microdermabrasion or medical-grade glycolic acid treatments to the treatment area within 2 weeks prior to participation.

Deep dermal scarring, thick sebaceous skin, or severe solar elastosis in the treatment area that may interfere with treatment or evaluation.

Intention to gain or lose ≥ 2 BMI units during the 12-month study period.

Known allergy or hypersensitivity to any component of the device or ultrasound coupling gel.

History of chronic drug or alcohol abuse or opioid dependence.

Recent aesthetic procedures to the lower face, submentum, or neck that may confound study outcomes (e.g., fillers, neurotoxins, lasers, threads, RF, ultrasound) within the protocol-specified washout period.

Participation in another clinical study involving an investigational device or drug within 30 days prior to treatment.

Pregnancy, breastfeeding, or plans to become pregnant during the study.

Any condition that, in the opinion of the investigator, would increase risk or interfere with study participation or data interpretation.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Laxity and Wrinkle Severity of the Lower Face and Neck | Baseline to 3 months post-treatment
  Clinical improvement in skin laxity, lines, and wrinkles of the lower face, submentum, and neck will be assessed by the Principal Investigator using the Global Aesthetic Improvement Scale (GAIS) and standardized 2D/3D photographs. The primary endpoint evaluates whether treatment with Ultherapy Prime results in a measurable improvement in lifting, tightening, and skin smoothness compared with baseline. GAIS scores range from "Very Much Improved" to "Worse," with higher ratings indicating greater aesthetic improvement.

SECONDARY OUTCOMES:
Change in Skin Laxity, Lines, and Wrinkle Severity at 6 and 12 Months | Baseline to 6 months, and Baseline to 12 months
  Evaluation of whether aesthetic improvement persists at 12 months using GAIS, photography, and patient satisfaction surveys to assess the duration of clinical benefit following a single MFU-V treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Levine, MD, Principal Investigator — Principal Investigator
Locations (1):
- The Levine Center for Plastic Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No